CLINICAL TRIAL: NCT05841108
Title: Effect of Task-oriented Training Assisted by Force Feedback Hand Rehabilitation Robot on Finger Function in Stroke Patients With Hemiplegia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Zhenlan li, department director, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20220101
Record Dates: First submitted 2023-02-14; First posted 2023-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Stroke
Keywords: Hand dysfunction; Force feedback hand rehabilitation robot; Task-oriented training; Neurorehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Device: force feedback rehabilitation robot (SEM™ Glove)
- control group (Active Comparator)
  Interventions: Other: assisted by a therapist

INTERVENTIONS:
Device: force feedback rehabilitation robot (SEM™ Glove) — In the experimental group, the therapists were asked to illustrate and demonstrate the motor points of the cylindrical grasping and spherical grasping movements, and the patients were instructed to imitate them with nonparalytic hand, while the latter patients wore SEM™ Glove were used for task-oriented training, such as inserting pegs, grasping a ball into a barrel, and drinking water exercises. The difficulty of task-oriented training can be adjusted according to the patient's actual condition, such as changing the shape, weight, size of the target or changing the distance, duration, and so on during training
  Other Names: SEM™ Glove
  Arms: experimental group
Other: assisted by a therapist — The control group received task-oriented training assisted by a therapist to complete the same task as the experimental group. Therapists need to instruct patients to try to grasp items and give appropriate assistance to guarantee their completion of the grasping task. If finger extension is weak, the therapist assists the patient in extension of the digits before grasping the items, and if the finger flexion angle does not meet the grasp function needs, it should assist in flexion finger movements
  Arms: control group

SUMMARY:
Over eighty percent of stroke patients experience finger-grasping dysfunction problems, compromising independence in daily life activities and quality of life. In routine training, task-oriented training is usually used for functional training of the hand, which may improve the finger grasping performance after stroke, whereby augmented therapy may lead to a better treatment outcome. Technology-supported training holds opportunities for increasing training intensity. However, most of the hand rehabilitation robots commonly used in the clinic are based on passive training mode and lacks the sensory feedback function of fingers, which is not conducive to patients completing more accurate grasping movements. The force feedback hand rehabilitation robot can make up for the above defects, but its clinical efficacy in stroke patients are not known to date. The aim of the present study was to investigate the effectiveness and added value of the force feedback hand rehabilitation robot combined with task-oriented training for stroke patients with hemiplegia.

ELIGIBILITY:
Inclusion Criteria:

* First-ever stroke
* Aged 20~80 years old
* Post-stroke time≤6 months
* Clinically diagnosed with a central paresis of the right arm/hand (Brunnstrom stage of the affected upper limb≥II, Brunnstrom stage of the affected hand II~V, Active flexion range of motion of the affected finger joint≥10°, MAS of affected upper limb and finger≤1+
* Sitting balance≥Level 2
* No serious depression and no visual impairment
* Cognitive and speech abilities sufficient to understand instructions and to provide informed consent

Exclusion Criteria:

* Severe additional neurological, orthopedic, or rheumatoid impairments before stroke which could interfere with task performance
* Sensory disturbance of fingers
* Severe joint pain caused by various reasons affects the functional activities of fingers
* Complicated with serious heart, lung, liver, kidney or infection
* Attending another study or therapy to improve arm-hand function

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-11-10 (Estimated); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer motor function assessment-upper limb finger motor part | Change from baseline Fugl-Meyer motor function assessment-upper limb finger motor part score at 4 weeks
  Fugl-meyer motor function assessment-upper limb (FMA-UL) has been found a reliable and valid test for the assessment of arm hand function in stroke patients. The maximum score of on the FMA-UL is 66 points. This study used FMA-UL finger motor part , with a total score of 14 points.

SECONDARY OUTCOMES:
Modified Ashworth scale (MAS) | Change from baseline Modified Ashworth scale outcome at 4 weeks
  The Modified Ashworth scale (MAS) was used to rate muscle tone/stiffness during passive movement of the flexors of the fingers. The scale ranges from '0 = normal','1','1+','2','3', and '4= worst'. Participants were assessed in all sessions using this 6-point ordinal scale for the hand treated in the study
Range of motion (ROM) | Change from baseline range of motion outcome at 4 weeks
  Range of motion (ROM) was measured with a goniometer. This study measures ROM of each finger, sum of five fingers flexion ROM, sum of five fingers extension ROM and total ROM of the five fingers. The ROM of each finger is the difference between the total ROM of each finger joint in the extension position and the total ROM of each finger joint in the flexion position. The sum of five finger flexion ROM is the sum of 14 finger joint flexion ROM. The sum of five finger extension ROM is the sum of 14 finger joint extension ROM. The total ROM of the five fingers is the difference between the total ROM of the extension position and the total ROM of the flexion position. The goniometer is used to measure the AROM of the affected hand first, and then the PROM.
grip strength | Change from baseline grip strength at 4 weeks
  Grip strength of the dominant hand was tested using an isometric hand dynamometer in the testing position recommended by American Society of Hand Therapists(ASHT). Participants gripped the dynamometer as hard as possible once without any jerking. The best score out of three consecutive trials was used for analyses. Sufficient time was allowed for the participants to recover from any fatigue related to grip testing
Brunnstrom recovery stages of hand (BRS-H) | Change from baseline brunnstrom recovery stages of hand at 4 weeks
  Brunnstrom recovery stages of hand (BRS-H) classifies the motor function into 6 levels based on recovery stages from a flaccid limb to near-normal and normal movement and coordination. Higher levels indicate better motor function. This study, the I-VI levels of the motor function were assigned with a score from 1 to 6.
Barthel index (BI) | Change from baseline barthel index at 4 weeks
  Barthel index contains 10 items and has a score range from 0 to 100, was used to assess activity and participation

CONTACTS AND LOCATIONS:
Locations (1):
- First hospital of Jilin University, Changchun, China

REFERENCES:
- [Derived] Li Y, Lian Y, Chen X, Zhang H, Xu G, Duan H, Xie X, Li Z. Effect of task-oriented training assisted by force feedback hand rehabilitation robot on finger grasping function in stroke patients with hemiplegia: a randomised controlled trial. J Neuroeng Rehabil. 2024 May 14;21(1):77. doi: 10.1186/s12984-024-01372-3. PMID 38745227